CLINICAL TRIAL: NCT02400424
Title: Multicenter Prospective Study of the Efficacy of Stereotactic Lung Radiation Therapy After Concomitant Radio-chemotherapy for Unresectable Stage III Non-small Cell Lung Carcinoma (NSCLC) With Peripheral Primary Tumor.
Brief Title: Study of the Efficacy of SBRT on Unresectable Peripheral Primary Tumor
Acronym: GFPC_01-14
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Approval of adjuvant durvalumab after RT-CT (not anticipated in the study design) and small number of stage III NSLCL patients with peripheral tumor accessible to SBRT
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFPC 01-14
Record Dates: First submitted 2015-03-11; First posted 2015-03-27 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Non-small-cell Lung Carcinoma
Keywords: Stereotactic lung radiation therapy; Radiochemotherapy; Unresectable stage III Non-Small Cell lung Carcinoma; Peripheral primary tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SBRT (Experimental): Study treatment = SBRT for peripheral primary tumor.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — 54 Gy in 3 fractions D1-D3-D5. SBRT should be started within 3 to 4 weeks after the end of radiochemotheray (RT-CT).
  Other Names: Stereotactic body radiation therapy

SUMMARY:
The purpose of this study is to evaluate the efficacy of stereotactic lung radiation therapy after concomitant radiochemotherapy for unresectable stage III non-small cell lung carcinoma (NSCLC) with peripheral primary tumor.

Evaluate in terms of local control rate at 6 months the addition of stereotactic radiotherapy after concurrent chemoradiotherapy in the treatment of mediastinal non-resectable stage III NSCLC having a peripheral primary tumor.

The number of patients required in this multicenter prospective study is 70.

This is a prospective, multicenter, non comparative and non randomized study.

DETAILED DESCRIPTION:
Stereotactic radiotherapy or SBRT (Body Stereotactic Radiation Therapy) allows to irradiate with high dose limited lesions size with a local control surrounding of 80-98% and with a low level of toxicity.

We propose to realize a classic concomitant RT-CT for mediastinal irradiation and combine this treatment with stereotactic RT for peripheral primary tumor.

The estimated inclusion period is approximately 3 years.

Follow-up duration for each patient is 2 years. The duration of the research is 5 years.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ Age ≤ 75 years
* PS ECOG 0 or 1
* Histologically proven NSCLC
* Unresectable stage III: T1 or T2 or T3 ≤ 5 cm AND N2 or N3 (only contralateral mediastinum or homolateral supraclavicular).
* Peripheral primary tumor ≥ 1 cm and ≤ 5 cm
* Possible concomitant chemoradiotherapy : 1 cure induction and 3 concomitant cycles of chemotherapy with cisplatin and Navelbine ® and 3D conformal radiotherapy delivering 66 Gy in 33 fractions to the mediastinal lymph node involvement without treating the peripheral tumor.
* Adequate biological parameters
* Forced expiratory volume (FEV) ≥1 liter or ≥ 30% of the theoretical value
* Patient covered by a health insurance scheme
* Signed informed consent

Exclusion Criteria:

* SCLC or large cell neuroendocrine carcinoma
* Metastatic disease
* Stage IVa
* Pregnant or breast-feeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-02; Primary Completion 2019-02-13 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Local control rate | 6 months after the end of SBRT
  According to RECIST v1.1

SECONDARY OUTCOMES:
Overall survival | From date of inclusion until the date of death from any cause, assessed up to 24 months after the end of SBRT
Progression-free survival | From date of inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months after the end of SBRT
Safety (adverse events, assessed using the NCI-CTCAE v4 grading scale) | Up to 2 years after the end of SBRT
  Incidence of adverse events, assessed using the NCI-CTCAE v4 grading scale

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle IM Martel Lafay, MD, Principal Investigator — Center Leon Berard
Locations (2):
- France (2):
  - Centre Leon Berard, Lyon
  - Hopital Nord-Ouest, Villefranche